CLINICAL TRIAL: NCT07159815
Title: Comparing the Health Benefits of Digital Home-based Resistance Exercise and Supervised On-site Resistance Exercise in Cancer Patients After Treatment - a 12 Week RCT.
Brief Title: REACT - Resistance Exercise After Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Stian Ellefsen, Professor, Inland Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR033
Record Dates: First submitted 2023-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The project is an assessor-blinded randomized controlled trial, where included participants will be randomized to either 12 weeks of digital home-based resistance exercise or the same program conducted in a studio under guidance of an instructor.
Who Masked: Outcomes Assessor
Masking Description: Assessment of all the outcomes will be performed in a blinded fashion by assessors/investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital home-based resistance exercise (Experimental): Participants in the digital group will need an e-mail and access to a pc and/or ipad at home. They will get access to a closed group on a digital platform, for participants in the project only. They will be asked to perform two pre-recorded resistance exercise sessions each week, for 12 weeks. Each session last for 40 minutes, and include 10 minutes of warm-up (ldynamic mobility and low impact), 25 minutes of resistance exercises (8-15 repetitions x 2-4 sets), and 5 minutes of cool-down and stretching. A total of 24 exercises will be performed over the period of 12 weeks.
  Interventions: Other: Digital follow-up; Behavioral: Resistance exercise
- On-site resistance exercise (Experimental): Participants in the on-site group will be asked to participate in resistance exercise on-site with instructor, two times a week for 12 weeks. They will follow the exact same exercise program as the digital group. Participants living around the Gjøvik area will have their exercise sessions at The Inland hospital Gjøvik (with physiotherapist and instructor supervising/mentoring the students), and for participants living around Lillehammer the exercise will be held at a medical clinic (with physiotherapist and instructor supervising/mentoring the students). A total of 24 exercises will be performed over the period of 12 weeks.
  Interventions: Other: On-site follow-up; Behavioral: Resistance exercise

INTERVENTIONS:
Other: Digital follow-up — See the arm/group description.
  Other Names: Cancer rehabilitation, digital follow-up
  Arms: Digital home-based resistance exercise
Other: On-site follow-up — See the arm/group description.
  Other Names: On-site cancer rehabilitation, on-site follow-up
  Arms: On-site resistance exercise
Behavioral: Resistance exercise — See the arm/group description.
  Other Names: Cancer rehabilitation

SUMMARY:
Resistance exercise has been shown to improve several important health variables after cancer and cancer related treatment, but unfortunately the adherence to resistance exercise is low. Typical reported exercise barriers are inconvenient location (e.g. long distance from home), exercise at an unfavorable time of the day, inadequate access to cancer-specific exercise and insufficient recommendations from healthcare providers. Thus, there is need for more research on resistance exercise with an alternative approach in cancer rehabilitation, that potentially can target a broad range of patients, despite their domicile. In Norway, the foundation "Active against cancer" has established exercise locations tareting cancer patients in several hospitals, and today they also offer digital home-based exercise sessions. Therefore, the overall research objectives are to compare the efficacy of 12 weeks digital, home-based resistance exercise program on cancer patients after treatment on functional, mental, and metabolic health, compared to the same program conducted in a studio under guidance of an instructor. The primary aim is to compare the effect on exercise adherence between digital home-based exercise program and on-site guided program on cancer patients after treatment. Secondary aims are to compare the two groups on several functional health outcomes, mental health outcomes and metabolic health markers.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and able to give informed consent
* Previously diagnosed with any form of cancer and completed systemic chemotherapy, immunotherapy or targeted therapies or local radiotherapy
* Have completed active cancer treatment not more than 12 months earlier or at present undergoing oral home-based treatment for stabilization or other treatments of disease or to prevent relapse
* Life expectancy of more than 12 months
* Digital opportunities at home: e.g axcess to pc, and/or ipad, email adress to log on the platform
* Able to understand Norwegian language

Exclusion Criteria:

* Co-morbidities prohibiting exercise according to protocol like serious cardic, pulmonary and other organ diseases
* Conditions caused by the cancer which prohibits exercise like previous major surgery, fractures, pain
* Still undergoing active cancer treatment that is expected to confer a high risk of bone marrow suppresion that would lead to infections, bleeding and/or severly reduced physical capacity
* Life expectancy of less than 12 months
* Reduced mental capacity and not able to give informed consent and follow the program
* Travelling distance more than 20 km from home or workplace to the two exercise locations (Gjøvik and/or Lillehammer) for patients who are candidates for randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Exercise adherence | From baseline to pre-test (0-12 weeks)
  Percentage of completed prescribed exercise sessions.

SECONDARY OUTCOMES:
Fatigue | From baseline to pre-test (0-12 weeks)
  Fatigue measured using "Chalder's Fatigue" questionnaire. This is 11 item questionnaire, where respondents first answer with a 1 or a 0 to indicate if the question apply to them or not, and then there is a Likert scale from 0 to 3 indicating each statement from "less than usual" to "much more than usual". The first part indicates the number of symptoms, and the other part the intensity of the symptoms. The global score can range from 0-33, where higher score indicates more fatigue.
Quality of life | From baseline to pre-test (0-12 weeks)
  Quality of life will be measured using the Short Form Health Survey (SF-36 questionnaire). SF-36 include 36 questions, covering eight domains of health. Each domain has a score being converted and pooled using a scoring key, indicating high or low quality of life. Likert scales and yes/no options are used in the questionnaire. The score in SF-36 are standardized in a two-step process by the SF-36v2 software, to obtain a scoring algoritm from 0-100. A higher score indicates better health state, and a score of 50 have been proposed as a normative value.
Cancer related quality of life | From baseline to pre-test (0-12 weeks)
  Cancer related quality of life will be measured using the European Organisation for Research and Treatment of Cancer Questionnaire (EORTC QLQ-C30 questionnaire), including five functional scales, three symptom scales, a global health status scale and six single items. All items range from 0 to 100, with a high scale score representing a higher response level, meaning a high score on the functional scale represents high level of functioning, a high score for the global health status represents high quality of life, but a high score on the symptom scale represents a high level of symptom.
Depression | From baseline to pre-test (0-12 weeks)
  Despression measured using the "Patient Health Questionnaire" (PHQ9). PHQ9 is a Likert scale where respondens score 0-4 on the nine items (ranging from "not at all" to "nearly every day". The total number of points are 27, and score 20-27 indicate severe depression. A total score from 1-4 indicate minimal depression, a score 5-9 indicate mild depression, score 10-14 indicate moderate depression and 15-19 indicate moderately severe depression.
Maximal muscle strength | From baseline to pre-test (0-12 weeks)
  Maximal muscle strength measured using one repetition maximum test (1RM) in leg press (Keiser) and leg extension (Humac)
Muscular endurance | From baseline to pre-test (0-12 weeks)
  Muscular endurance measured using correctly performed number of repetitions with 70% of 1RM in leg press (Keiser) and leg extrension (Humac)
Functional fitness, six minutes step test | From baseline to pre-test (0-12 weeks)
  Functional fitness measured using the "six minutes step" test
Functional fitness, sit to stand test | From baseline to pre-test (0-12 weeks)
  Functional fitness measured using the "sit to stand test" (30 sec)
Muscle mass, DXA scan | From baseline to pre-test (0-12 weeks)
  Muscle mass measured using the whole-body DXA scan
Visceral fat mass, DXA scan | From baseline to pre-test (0-12 weeks)
  Visceral fat mass measured using the whole-body DXA scan
Muscle mass, ultrasound | From baseline to pre-test (0-12 weeks)
  Muscle mass measured using ultrasound to detect muscle thivkness of m.vastus lateralis
Lipoprotein profile (subclasses of LDL, HDL) | From baseline to pre-test (0-12 weeks)
  Number of participants with improvements in lipoprotein profile (subclasses of LDL, HDL) measured taking venous blood samples
Blood pressure at rest | From baseline to pre-test (0-12 weeks)
  Both systolic and diastolic blood pressure at rest measured using automated upper-arm blood pressure cuff
Fasting blood glucose | From baseline to pre-test (0-12 weeks)
  Number of participants with improvement in fasting blood glucose measured in serum
Hemoglobin glycosylation (HbA1c) | From baseline to pre-test (0-12 weeks)
  Number of participants with improvements in long-term glucose levels measured as hemoglobin glycosylation of the metabolic syndrome such as waist circumference, blood pressure at rest, lipid profile (hemoglobin glycosylation (HbA1c) and fasting blood glucose
Waist circumference | From baseline to pre-test (0-12 weeks)
  Number of participants with reduction in circumference of the waist measured using measuring tape.
Glucose tolerance (c-peptide) | From baseline to pre-test (0-12 weeks)
  Oral glucose tolerance test (c-peptide) using venous blood samples
Glucose tolerance (glucose) | From baseline to pre-test (0-12 weeks)
  Oral glucose tolerance test (glucose) using venous blood samples
Triglycerides | From baseline to pre-test (0-12 weeks)
  Number of participants with improvements in triglycerides measured using venous blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: No